CLINICAL TRIAL: NCT02232997
Title: The Optimal Hydration With Sodium Chloride in High Risk Patients Undergoing Coronary Angiography, Reduction of Risk of Contrast-associated Acute Kidney Injury After Cardiac Catheterization 2 (TIME RESCIND 2) Study
Brief Title: Simplified Rapid Hydration in Preventing CA-AKI Among Patients With Chronic Kidney Disease
Acronym: TIME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guangdong Provincial People's Hospital (Other)
Collaborators: Peking University First Hospital (Other); Fudan University (Other); The General Hospital of Northern Theater Command (Other); Xiamen Cardiovascular Hospital, Xiamen University (Other); First Affiliated Hospital of Guangxi Medical University (Other); Sichuan Provincial People's Hospital (Other); Wuhan Asia Heart Hospital (Other); West China Hospital (Other); Jining Medical University (Other); The First Affiliated Hospital of Zhengzhou University (Other); Fujian Provincial Hospital (Other); First Affiliated Hospital, Sun Yat-Sen University (Other); Fuling Central Hospital of Chongqing City (Other); Second Xiangya Hospital of Central South University (Other); People's Hospital of Guangxi Zhuang Autonomous Region (Other); Maoming People's Hospital (Other); Xijing Hospital (Other); Beijing Friendship Hospital (Other); Tangshan Gongren Hospital (Other); Xuzhou Central Hospital (Other); Southern Medical University, China (Other)
Responsible Party: Principal Investigator, Jiyan Chen, MD, Guangdong Provincial People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CSC20140818; CSC20140818 (Other: Chinese Society of Cardiology)
Record Dates: First submitted 2014-09-01; First posted 2014-09-08 (Estimated); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: Chronic Kidney Disease
Keywords: Contrast-associated acute kidney injury; Coronary angiography; Chronic kidney disease; Intravenous hydration
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard Hydration (Active Comparator): Standard long-term hydration, i.e. hydrated with normal saline 12 hours before and 12 hours after coronary intervention at a rate of 1 ml/kg/h
  Interventions: Other: Standard Hydration
- Simplified Hydration (Active Comparator): Rapid short-term hydration, i.e. hydrated with normal saline from 1 hour before to 4 hours after coronary intervention at a rate of 3 ml/kg/h
  Interventions: Other: Simplified Hydration

INTERVENTIONS:
Other: Standard Hydration — Sodium chloride hydration was set between 12 hours before coronary intervention (before contrast exposure during coronary angiography), continued during procedure, and 12 hours after procedure at 1 ml/kg/h (0.5 ml/kg/h For patients with congestive heart failure, New York Heart Association class>II, or LVEF < 35%). For patients weighing more than 80 kg, bolus and infusion rates are limited to calculated values for patients weighing 80 kg
  Other Names: The control hydration group
  Arms: Standard Hydration
Other: Simplified Hydration — Hydration with sodium chloride was set 1 hour before procedure (before contrast exposure during coronary angiography), continued during procedure, and 4 hours after procedure at 3ml/kg/h (1.5ml/kg/h For patients with congestive heart failure, New York Heart Association class>II, or LVEF <35%). For patients weighing more than 80 kg, bolus and infusion rates are limited to those calculated for patients weighing 80 kg.
  Other Names: The simple hydration group
  Arms: Simplified Hydration

SUMMARY:
No well-defined protocols exist to guide fluid administration for prevention of contrast-associated acute kidney injury in high risk patients. The investigators will compare long term hydration at routine speed(12h before and after procedure at 1ml/kg/h) with short term hydration at high speed(1h before and 4h after procedure at 3ml/kg/h) to verify our hypothesis that the short term hydration may not be inferior to the long one.

DETAILED DESCRIPTION:
No well-defined protocols exist to guide fluid administration for prevention of contrast-associated acute kidney injury in high risk patients undergoing coronary angiography. Long term hydration at routine speed(12h before and after procedure at 1ml/kg/h), as the most recommended adequate hydration, has been carried out to prevent contrast-associated acute kidney injury in lots of clinical trials. Base on the data in the POSEIDON randomized controlled trial with hemodynamic-guided fluid administration, short term hydration at high speed(1h before and 4h after procedure at 3ml/kg/h) may not be inferior to the classic long term hydration, the speed should be reduced half of the intended speed in all the patients. We hypothesized short term hydration may not be inferior to the long one to reduced significantly the hospital stay and healthy cost.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age;
* Written informed consent;
* Candidates scheduled for coronary intervention (angiography and/or coronary intervention);
* Patients with chronic renal insufficiency, the baseline estimated glomerular filtration rate (eGFR) was 15-60 mL/min / 1.73 m²
* At least one risk factor (age>75 years, medical history of diabetes mellitus or hypertension, congestive heart failure [NYHA class >II or history of acute pulmonary edema]);

Exclusion Criteria:

* End-stage renal failure or heart/renal transplantation;
* History of exposure to contrast medium or acute infectious diseases within 48 hours prior to the procedure;
* Acute decompensated heart failure;
* Left ventricular thrombus;
* Allergy to contrast agent;
* Pregnancy or lactation;
* Malignant tumour or life expectancy <1 year;
* Pre-procedural receipt of NSAIDs (except Asprin), aminoglycosides, cyclosporine or cisplatin in the past 48 h;
* Severe valve disease or elective undergoing surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1002 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2021-12 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
Contrast-associated acute kidney injury a | 72 hours
  Defined as ≥25% or 0.5 mg/dL absolute increase in serum creatinine from baseline during the first 48-72 hours after the procedure

SECONDARY OUTCOMES:
Number of Participants with Acute heart failure | post-procedural during hospitalization, an average of 3 days
  Defined as signs/symptoms of heart congestion and/or hypoperfusion by physical examination and auxiliary examination such as ECG, chest X-ray, laboratory assessment (biomarkers and echocardiography)
Contrast-associated acute kidney injury b | 72 hours
  Defined as ≥0.5 mg/dL increase in serum creatinine from baseline during the first 48-72 hours after the procedure
Contrast-associated acute kidney injury c | 24 hours
  Defined as ≥10% increase in serum cystatin c from baseline during the first 24 hours after the procedure
Contrast-associated acute kidney injury d | 48 hours
  Defined as ≥50% or 0.3 mg/dL increase in serum creatinine from baseline during the first 48 hours after the procedure
Contrast-associated acute kidney injury e | 24 hours
  Defined as ≥0.3mg/dl increase in serum cystatin c from baseline during the first 24 hours after the procedure
Major adverse clinical events | 1 year
  Including all-cause mortality, renal replacement therapy, nonfatal myocardial infarction, acute pulmonary edema, stroke, rehospitalization, bleeding
Change in eGFR a | 72 hours
  Change in eGFR within 48-72 hours after procedure (calculated according to the simplified MDRD formula)
Change in eGFR b | 72 hours
  Change in eGFR within 48-72 hours after procedure (calculated according to the Cysc)
Contrast-induced persistence kidney injury | 3 months
  Defined as residual impairment of renal function indicated by a >25% reduction in creatinine clearance in comparison with the baseline value or dialysis requirement at 3 months
Length of stay | an average of 7 days
  Total length of hospital stay
Total hospitalization costs | an average of 7 days
  Hospitalization expenses during hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Jiyan Chen, MD, Study Chair — Guangdong Cardiovascular Institute, Guangdong Provincial People's Hospital; Yong Liu, MD, Study Director — Guangdong Cardiovascular Institute, Guangdong Provincial People's Hospital; Yong Huo, MD, Principal Investigator — Peking University First Hospital; Junbo Ge, MD, Principal Investigator — Fudan University; Pingyan Chen, MS, Principal Investigator — Southern Medical University
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, Guangdong, China